CLINICAL TRIAL: NCT03245554
Title: Clinical Research on Teratment of Gastrointestinal Cancer in the Preoperative by Propranolol
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yijing He, Associate Professor, Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017 PROP/CSU/GC
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal Cancer; Propranolol
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- placebo and propranolol (Experimental): We used propranolol and placebo as an control drug to treat with patients.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — 0 or 1 were generated by using Random software. The patient entered the placebo group if number was 0; if the random number generated was 1, then entered the propranolol group.
  Other Names: placebo

SUMMARY:
To research the effect of propranolol on the proliferation and apoptosis of gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. patients with gastric adenocarcinoma and colon cancer were diagnosed by histology and cytology, and there was a clear metastasis (TxNxM0);
2. without any prior treatment (including surgery or radiotherapy and chemotherapy) in the I-III period, no distant metastasis, suitable for patients with surgical resection of the tumor.
3. the age range of the patients is 18-60;
4. systolic pressure 100-140mmHg; heart rate >60bpm;
5. the patient's survival time should be longer than 3 months;
6. without previous cardiovascular and cerebrovascular diseases, the atrioventricular block was excluded by the 24 hour dynamic electrocardiogram;
7. ECOG score of 2 (that means the patient's bed time is less than 50%); Karnofsky score of 60% (that means patients have the basic activities and self-care ability);
8. the basic biochemical examination results of patients with normal: white blood cell 3000/ul; neutrophil 1500/ul 100000/ul; platelet count; total bilirubin < 1.5 x ULN; AST / ALT 2.5 x ULN without liver metastasis; < 5 x ULN liver metastasis; creatinine clearance rate of 1.5 x ULN;
9. have the ability to understand and sign informed consent.

Exclusion Criteria:

1. pregnant or lactating women;
2. patients with severe heart disease, kidney disease, metabolic disorders, bronchial asthma, cardiogenic shock, heart block (II-III degree atrioventricular block), or severe acute heart failure, sinus bradycardia.
3. patients with epilepsy or psychotropic drugs and sedatives;
4. patients with brain metastasis and bone marrow metastasis;
5. participants in clinical trials of other drugs within 4 weeks;
6. patients with a history of anaphylaxis with propranolol;
7. patients treated with trastuzumab;
8. patients with or reactive immunodeficiency, such as those with HIV infection;
9. the uncontrollable situation in the group during the period (but not limited to these cases): according to the experimental scheme of medication, severe infection, due to mental illness or other social factors lead to the compliance requirements of patients;
10. patients with atrioventricular block should be discontinued immediately and quit;
11. the researchers believe there may be any increase in the risk of the subject or any interference with clinical trials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Tumor size will be measured. | Our experiment completed after patients took medicine for one week.
  We used CT and Ki67 to confirm that the drug's affection.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Clinical Pharmacology, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided